CLINICAL TRIAL: NCT04343235
Title: Postpartum Management of Gestational Hypertensive Disorders Using Furosemide: A Randomized Controlled Trial
Brief Title: Postpartum Management of Gestational Hypertensive Disorders Using Furosemide
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Challenges with enrollment; primary investigator left the institution
Sponsor: Wright State University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 06784
Record Dates: First submitted 2019-10-28; First posted 2020-04-13 (Actual); Results first posted 2023-10-23 (Actual); Last update posted 2023-10-23 (Actual); Status verified 2023-09

CONDITIONS: Hypertension, Pregnancy-Induced
Keywords: pregnancy induced hypertension; preeclampsia; furosemide
MeSH Terms: conditions — Hypertension, Pregnancy-Induced; Pre-Eclampsia | interventions — Furosemide; Labetalol

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Masking Description: randomized open label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- labetalol + furosemide (Experimental): labetalol + furosemide
  Interventions: Drug: furosemide; Drug: labetalol
- labetalol only (Active Comparator): labetalol only
  Interventions: Drug: labetalol

INTERVENTIONS:
Drug: furosemide — five day course of furosemide 20mg QD
  Other Names: lasix
  Arms: labetalol + furosemide
Drug: labetalol — 200mg labetalol BID
  Other Names: trandate

SUMMARY:
* The main purpose of this study is to learn if incorporating a loop diuretic such as furosemide along with labetalol in the routine management of postpartum gestational hypertensive disorders could lower the need for additional anti-hypertensive agents to control blood pressures, improve blood pressures (as measured by systolic blood pressure, diastolic blood pressure and mean arterial blood pressures), shorten hospital stays and decrease readmissions for patients with gestational hypertensive disorders.
* Based on a study by Veena et al1, there is reason to believe that the addition of furosemide to other anti-hypertensives may help decrease the need to add or increase the dose of medication to control blood pressures. There may be potential to shorten hospital stays and decrease readmissions, as well. Collecting data will be done using a prospective, randomized 1:1 controlled study assigning postpartum patients with a gestational hypertensive diagnosis to either labetalol alone or labetalol plus furosemide.
* The study will be performed in the postpartum wing of Miami Valley Hospital Main Campus and would use patients who have consented to participate in the study with enrollees coming from the OB Staff population.

DETAILED DESCRIPTION:
Background and Literature Review

* There have been four documented studies investigating loop diuretics in the management of postpartum hypertensive disorders- Matthews et al2, Ascarelli et al3, Amorim et al4, and Veena et al. Of these studies, only Amorim and Veena were able to show statistical significance on any parameters. Amorim was able to show that there was an improvement of SBP, DBP and MAP, but the research was only presented as an abstract at a conference and not published, thereby making it impossible to draw any conclusions or practice guidelines. Veena demonstrated that by using furosemide and nifedipine in combination, the need for additional antihypertensive medication in severe pre-eclampsia in the postpartum period was reduced when compared to nifedipine alone.
* A systematic review5 of postpartum hypertensive disorder management suggested that there was insufficient data to recommend any single pharmacological intervention at this time in the management of gestational hypertensive disorders. The review emphasized the need for further studies to be conducted to help guide management of patients affected by gestational hypertensive disorders in the future.

Objectives

● Main Question

* Does the use of furosemide plus labetalol improve blood pressures in the postpartum period of patients with gestational hypertensive disorders versus labetalol alone?
* Primary

  ■ Will there be a requirement to escalate antihypertensive therapy to control blood pressures
* Secondary

  * Improvement of gestational hypertensive disorders by measurement of systolic blood pressure, diastolic blood pressure and mean arterial pressure
  * Shortened hospital stay in patients with hypertensive disorders
  * Breastfeeding status at 1 week postpartum visit in mothers planning to breastfeed
  * Readmission for postpartum hypertensive disorders

Significance to patient, institution, and profession

* As a referral center and being the region's leader, Miami Valley is very accustomed to accepting transfers of high acuity patients often times with hypertensive disorders being the root cause of the transport
* The majority of the OB staff population being served at Miami Valley Hospital is African American. According to Myatt6, the incidence of pre-eclampsia in the African American population is greater than double the Caucasian population (11% to 5%) thereby making this study very applicable to the patient population served at Miami Valley Hospital.
* With the construct of the study, costs abe kept low by utilizing already established resources and practices (blood pressure cuffs, nurses, routine one week blood pressure checks) while only adding on the unit cost of furosemide.
* If treatment with labetalol and furosemide is found to be useful, it would be not only a very inexpensive, cost effective way of improving patient outcomes and possibly decreasing lengths of stay stateside, but in improving global practice in places that are lacking in resources privy to first world countries.

Methods

* The study would be designed as:

  * A prospective randomized 1:1 controlled trial including postpartum women with gestational hypertension or preeclampsia
  * Patients with chronic hypertension would be excluded from the study
  * One arm receiving 200mg labetalol BID alone on PPD#1 or 24 hours after magnesium sulfate
  * One arm receiving 200mg labetalol BID and a five day course of furosemide 20mg QD on PPD#1 or 24 hours after magnesium sulfate
  * Recording any occurrence when an increased amount of labetalol is needed to maintain blood pressures below 150 SBP and/or 100 DBP per ACOG recommendations.7

    ■ In the event of persistently elevated blood pressures, labetalol will be increased to 400mg TID and escalated to 600mg TID and finally 800mg TID as indicated
  * Measurement of blood pressure every four hours after administration until patient discharge
  * Measurement of urine output every 12 hours until discharge
  * Compare average systolic, diastolic and mean arterial pressures between the two groups during admission and at one week postpartum
* Data will be collected using the OB Staff population at Miami Valley Hospital Main Campus.
* The research will be analyzed and interpreted by the research team conducting the study.
* Potential difficulties and limitations include compliance concerns of mandatory one week blood pressure follow up appointment.
* Using the Veena et al paper as a frame of reference, a sample size of 140 divided evenly across the two treatment arms would achieve statistical significance in determining the need to escalate anti-hypertensive therapy.
* The unit cost of one tablet of labetalol 200mg and furosemide 20mg is currently $0.32 and $1.23, respectively. 8,9
* The study would use already readily available automated blood pressure cuff machines on the postpartum wing.

ELIGIBILITY:
Inclusion Criteria:

* Postpartum women delivering at Miami Valley Hospital
* Diagnosis of gestational hypertension or preeclampsia
* Able to provide written informed consent

Exclusion Criteria:

* Diagnosis of chronic hypertension
* Allergy to study medications
* Unable to understand English

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Female
Enrollment: 13 (Actual)
Dates: Start 2020-05-01 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sheela Barhan, MD, Principal Investigator — Wright State University
Locations (1):
- Miami Valley Hospital, Dayton, Ohio, United States

IPD SHARING:
Plan to Share IPD: No
Data will be shared on a case by case basis

REFERENCES:
- [Background] Veena P, Perivela L, Raghavan SS. Furosemide in postpartum management of severe preeclampsia: A randomized controlled trial. Hypertens Pregnancy. 2017 Feb;36(1):84-89. doi: 10.1080/10641955.2016.1239735. Epub 2016 Nov 11. PMID 27835048
- [Background] Matthews G, Gornall R, Saunders NJ. A randomised placebo controlled trial of loop diuretics in moderate/severe pre-eclampsia, following delivery. J Obstet Gynaecol. 1997 Jan;17(1):30-2. doi: 10.1080/01443619750114040. PMID 15511760
- [Background] Ascarelli MH, Johnson V, McCreary H, Cushman J, May WL, Martin JN Jr. Postpartum preeclampsia management with furosemide: a randomized clinical trial. Obstet Gynecol. 2005 Jan;105(1):29-33. doi: 10.1097/01.AOG.0000148270.53433.66. PMID 15625138
- [Background] Cairns AE, Pealing L, Duffy JMN, Roberts N, Tucker KL, Leeson P, MacKillop LH, McManus RJ. Postpartum management of hypertensive disorders of pregnancy: a systematic review. BMJ Open. 2017 Nov 28;7(11):e018696. doi: 10.1136/bmjopen-2017-018696. PMID 29187414
- [Background] Myatt L, Clifton RG, Roberts JM, Spong CY, Hauth JC, Varner MW, Thorp JM Jr, Mercer BM, Peaceman AM, Ramin SM, Carpenter MW, Iams JD, Sciscione A, Harper M, Tolosa JE, Saade G, Sorokin Y, Anderson GD; Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) Maternal-Fetal Medicine Units (MFMU) Network. First-trimester prediction of preeclampsia in nulliparous women at low risk. Obstet Gynecol. 2012 Jun;119(6):1234-42. doi: 10.1097/AOG.0b013e3182571669. PMID 22617589
- [Background] Hypertension in pregnancy. Report of the American College of Obstetricians and Gynecologists' Task Force on Hypertension in Pregnancy. Obstet Gynecol. 2013 Nov;122(5):1122-1131. doi: 10.1097/01.AOG.0000437382.03963.88. No abstract available. PMID 24150027

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Labetalol + Furosemide | Labetalol Only
Started | 6 | 7
Completed | 3 | 5
Not Completed | 3 | 2
Not completed — Lost to Follow-up | 3 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Labetalol + Furosemide | Labetalol Only | Total
Number analyzed (Participants) | 6 | 7 | 13
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 6 | 7 | 13
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 28.0 (2.7) | 27.0 (5.4) | 27.5 (4.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 7 | 13
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 6 | 6 | 12
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 3 | 6
  White | 3 | 4 | 7
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 6 | 7 | 13

OUTCOME MEASURES:

1. Primary Outcome: Change of Dose for Antihypertensive Therapy
Description: number of patients who require a change in the dose of labetalol to control BP
Time Frame: Change in dose of hypertensive therapy from randomization until hospital discharge (up to 7 days)
Measure: Count of Participants; unit: Participants
Arm/Group | Labetalol + Furosemide | Labetalol Only
Number analyzed (Participants) | 6 | 7
Participants | 3 | 0
Statistical Analysis 1: Comparison: Labetalol + Furosemide vs Labetalol Only; Test type: Superiority; p = 0.21, Fisher Exact

2. Secondary Outcome: Change of Gestational Hypertensive Disorder Symptoms (Systolic BP)
Description: average systolic blood pressure reading on Day 0, Day 1, and Day 2
Time Frame: Average systolic blood pressure for Day 0, Day 1, and Day 2
Measure: Mean (Standard Deviation); unit: mm of mercury
Arm/Group | Labetalol + Furosemide | Labetalol Only
Number analyzed (Participants) | 4 | 7
mm of mercury
  Day 0 | 138.4 (11.2) | 138.1 (9.4)
  Day 1 | 134.9 (5.4) | 138.2 (8.5)
  Day 2 | 135.2 (13.7) | 136.7 (6.0)
Statistical Analysis 1: Comparison: Labetalol + Furosemide vs Labetalol Only; Test type: Superiority; p = 0.70, ANOVA — Main effect for Randomization group

3. Secondary Outcome: Change of Gestational Hypertensive Disorder Symptoms (Mean Arterial Pressure)
Description: average mean arterial pressure reading on Day 0, Day 1, and Day 2
Time Frame: Average mean arterial pressure on Day 0, Day 1, and Day 2
Measure: Mean (Standard Deviation); unit: mm of mercury
Arm/Group | Labetalol + Furosemide | Labetalol Only
Number analyzed (Participants) | 4 | 7
mm of mercury
  Day 0 | 102.4 (10.7) | 100.0 (9.2)
  Day 1 | 99.5 (4.7) | 100.1 (7.7)
  Day 2 | 98.0 (8.7) | 96.0 (6.3)
Statistical Analysis 1: Comparison: Labetalol + Furosemide vs Labetalol Only; Test type: Superiority; p = 0.77, ANOVA; Main effect for randomization group

4. Secondary Outcome: Change of Gestational Hypertensive Disorder Symptoms (Diastolic BP)
Description: average diastolic blood pressure reading on Day 0, Day 1, and Day 2
Time Frame: Average diastolic blood pressure on Day 0, Day 1, and Day 2
Measure: Mean (Standard Deviation); unit: mm of mercury
Arm/Group | Labetalol + Furosemide | Labetalol Only
Number analyzed (Participants) | 4 | 7
mm of mercury
  Day 0 | 84.1 (11.8) | 80.1 (10.4)
  Day 1 | 81.8 (4.5) | 80.7 (8.4)
  Day 2 | 78.8 (7.1) | 75.5 (7.9)
Statistical Analysis 1: Comparison: Labetalol + Furosemide vs Labetalol Only; Test type: Superiority; p = 0.54, ANOVA; Main effect for randomization group

5. Secondary Outcome: Hospital Length of Stay
Description: days in hospital after delivery
Time Frame: Number of days of hospital stay from randomization to discharge
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Labetalol + Furosemide | Labetalol Only
Number analyzed (Participants) | 6 | 7
days | 3.5 (1.3) | 4.3 (1.8)
Statistical Analysis 1: Comparison: Labetalol + Furosemide vs Labetalol Only; Test type: Superiority; p = 0.47, t-test, 2 sided; Mean Difference (Final Values) = .79, 95% CI 2-sided [-1.5 to 3.1], Standard Error of Mean 1.0

6. Secondary Outcome: Breastfeeding Status
Description: breastfeeding continuation after discharge
Time Frame: at 1 week postpartum visit
Measure: Count of Participants; unit: Participants
Arm/Group | Labetalol + Furosemide | Labetalol Only
Number analyzed (Participants) | 4 | 6
Participants | 1 | 3
Statistical Analysis 1: Comparison: Labetalol + Furosemide vs Labetalol Only; Test type: Superiority; p = 0.57, Fisher Exact

7. Secondary Outcome: Hospital Readmission
Description: readmission for hypertension management
Time Frame: up to 14 days after discharge
Measure: Count of Participants; unit: Participants
Arm/Group | Labetalol + Furosemide | Labetalol Only
Number analyzed (Participants) | 6 | 7
Participants | 1 | 2
Statistical Analysis 1: Comparison: Labetalol + Furosemide vs Labetalol Only; Test type: Superiority; p > 0.99, Fisher Exact

ADVERSE EVENTS:
Time Frame: 2 weeks
Description: Adverse events were used according to the clinicaltrials.gov definitions.
Arm/Group | Labetalol + Furosemide | Labetalol Only
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/7
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/7
Other Adverse Events (participants affected / at risk) | 0/6 | 0/7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2020-01-09): https://cdn.clinicaltrials.gov/large-docs/35/NCT04343235/Prot_000.pdf
  • Statistical Analysis Plan (2020-01-09): https://cdn.clinicaltrials.gov/large-docs/35/NCT04343235/SAP_003.pdf
  • Informed Consent Form (2022-01-10): https://cdn.clinicaltrials.gov/large-docs/35/NCT04343235/ICF_002.pdf